CLINICAL TRIAL: NCT06417996
Title: Postoperative Digital Care Home Monitoring
Brief Title: Biobeat Digital Home Monitoring Feasibility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Richard Malthaner, Chair/Head, Thoracic Surgery, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Digital Home Monitoring
Record Dates: First submitted 2024-02-21; First posted 2024-05-16 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Thoracic Surgery; Home Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will not be monitored with continuity of care.
- Digital Group (Experimental): At the time of hospital discharge, the control group will be discharged without receipt of home monitoring, and the intervention group will receive a home monitoring kit with (NIBP (non-invasive blood pressure) and SPO2 (pulse oximetry) with instructions on how to use these devices. Patients in the intervention groups will receive digital communication for four weeks and have their NIBP, HR (heart rate), SPO2 and pain scores evaluated twice a day for two weeks.
  Interventions: Other: Digital Group

INTERVENTIONS:
Other: Digital Group — Once patients are ready for discharge, patients in the digital group will be sent home with the Biobeat digital monitoring kit with written & oral instructions on how it will be used in maintaining continuity of care which will track ECG (electrocardiogram), HR, NIBP, SPO2, and pain scores. A continuous recording and two-lead ECG patch will be applied and activated at the time of discharge to identify any paroxysmal atrial fibrillation.
  Arms: Digital Group

SUMMARY:
To assess the feasibility of evaluating postoperative home monitoring with Biobeat digital monitoring. The investigators hypothesize that the Biobeat digital home monitoring platform will lead to a decrease in unplanned visits to the ED (Emergency Department). In addition, patients' quality of life is postulated to be improved compared to patients receiving the current standard of care without home monitoring.

DETAILED DESCRIPTION:
This trial will be a single centre, parallel arm, randomized controlled feasibility trial. The investigators will evaluate postoperative home monitoring with the Biobeat digital monitoring and two-way communication through the digital portal for 4 weeks post-operatively to the standard of care (no digital monitoring) in thoracic surgery patients undergoing elective thoracic surgical procedures. The investigators will assess whether conducting a larger randomized trial of digital home monitoring vs. standard of care is feasible in terms of recruitment, data collection and logistics.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing to provide informed consent
* Wi-fi or cellular connectivity at the patient's home
* Patient undergoing elective lung cancer surgery
* Patient familiar/comfortable with the use of technology such as online banking.

Exclusion Criteria:

- Patients who are not comfortable with the use of technology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess whether conducting a larger randomized trial of digital home monitoring vs. standard of care is feasible in terms of recruitment, data collection and logistics. | 365 days
  The trial will be deemed feasible if >/= 60% of eligible patients are recruited, >/= 80% of data is collected, and </= 20% of patients are lost to follow-up.

SECONDARY OUTCOMES:
Number of ED Visits | 30 days from discharge
  Number of ED visits
Readmission Rates | 30 days from discharge
  Number of readmissions

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No